CLINICAL TRIAL: NCT00775814
Title: Double-blind, Randomized Trial to Investigate the Antihypertensive and Metabolic Effects of Candesartan in Insulin-resistant Obese Patients With a Hypertension Not Adequately Controlled by Previous ß-blocker or Calcium Channel Blocker
Brief Title: Efficacy of Candesartan on Reducing Blood Pressure in Insulin-Resistant, Obese Patients With Hypertension.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BLO K025; 2006-001998-25 (EudraCT Number); D-CAN-545 (Other: Takeda ID); U1111-1113-9336 (Registry Identifier: WHO)
Record Dates: First submitted 2008-10-16; First posted 2008-10-20 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Obesity; Hypertension
Keywords: Hypertension; Drug Therapy; Blood Pressure; Insulin, Resistant
MeSH Terms: conditions — Obesity; Hypertension; Insulin Resistance | interventions — candesartan; Hydrochlorothiazide; candesartan cilexetil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Candesartan + Hydrochlorothiazide QD (Experimental)
  Interventions: Drug: Candesartan and Hydrochlorothiazide
- Hydrochlorothiazide QD (Active Comparator)
  Interventions: Drug: Hydrochlorothiazide (HCT)

INTERVENTIONS:
Drug: Candesartan and Hydrochlorothiazide — Candesartan 8 mg, tablets, orally, once daily and hydrochlorothiazide 12.5 mg, tablets, orally, once daily for 2 weeks; increased to Candesartan 16 mg, tablets, orally, once daily and hydrochlorothiazide 12.5 mg, tablets, orally, once daily for up to 24 weeks.
  Other Names: BLOPRESS PLUS®
  Arms: Candesartan + Hydrochlorothiazide QD
Drug: Hydrochlorothiazide (HCT) — Candesartan placebo-matching tablets and hydrochlorothiazide 12.5 mg, tablets, orally, once daily for up to 24 weeks.
  Arms: Hydrochlorothiazide QD

SUMMARY:
The purpose of this study is to determine the efficacy of candesartan, once daily (QD), combined with hydrochlorothiazide to lower blood pressure in insulin-resistant, obese patients with hypertension.

DETAILED DESCRIPTION:
Abdominal obesity is a major risk factor for insulin resistance and the development of type 2 diabetes. It is associated with sodium retention, left ventricular hypertrophy and elevated markers of inflammation and is an important predictor of cardiovascular morbidity and mortality. Activation of the sympathetic nervous system and the renin angiotensin aldosterone system are both involved in the development of hypertension in obese individuals. Hypertension in obese individuals is often associated with dyslipidemia, hyperinsulinaemia and impaired glucose tolerance.

In order to decrease the cardiovascular risk of obese hypertensive patients, therapy should not only be directed to lowering blood pressure values but also to improvement of their metabolic situation. As it is possible that antihypertensive treatment based on an angiotensin receptor antagonist (like candesartan) might be superior to beta-blocker or calcium channel blocker therapy in preventing diabetes, a combination of candesartan with already existing insufficiently effective beta-blocker or calcium channel blocker therapy will be used in this study.

ELIGIBILITY:
Inclusion Criteria:

* Has an Abdominal obesity with a waist circumference greater than 102 cm (men) and greater than 88 cm (women).
* Has a body mass index greater than 30 kg/m^2.
* Has hypertension not adequately controlled (seated diastolic blood pressure greater than 95 mmHg and less than or equal to 110 mmHg as median value of three readings) by monotherapy with either beta-blocker or calcium channel blocker.
* Has a Homeostasis Model Assessment Insulin Resistance index greater than 3.99.
* Has hyperlipidemia with fasting levels for total cholesterol greater than 250 mg/dL (6.45 mmol/L) or low-density lipoprotein cholesterol greater than 160 mg/dL (4.13 mmol/L) or triglycerides greater than 250 mg/dL (2.82 mmol/L).

Exclusion Criteria:

* Existing Hydrochlorothiazide therapy at start of study.
* Diabetes mellitus type 1 or 2 [known or newly detected (Screening: fasting plasma glucose greater than 7.0 mmol/L)].
* Chronic renal impairment or S-creatinine greater than or equal to 1.8 mg/dL.
* Presence of single kidney or state after kidney transplantation or known bilateral renal artery stenosis or interventional treatment for renal artery stenosis in the last year.
* Hyperkalemia (potassium greater than 5.5 mmol/L).
* Known electrolyte imbalance, e.g. hypocalcaemia or hypokalemia resistant to treatment.
* Nephrotic syndrome.
* Thyroid dysfunction.
* Primary or secondary hyperaldosteronism.
* Cushing syndrome.
* Known or suspected familial hypercholesterolemia.
* Severe hepatic impairment (cholestasis (bilirubin greater than 2.0 mg/dL) or alanine aminotransferase and/or aspartate aminotransferase greater than 3 times the upper limit of normal and/or γ-glutamyl transpeptidase greater than 5 times the upper limit of normal).
* History of chronic heart failure.
* History of overt coronary heart disease.
* History of silent myocardial infarction.
* Hemodynamically relevant stenosis of the mitral and/or aortic valve.
* History of stroke.
* Stage 3 hypertension (systolic blood pressure greater than 180 mmHg or diastolic blood pressure greater than 110 mmHg).
* Angiotensin converting enzyme inhibitor or angiotensin receptor blocker therapy in the previous 4 weeks.
* Lipid-lowering therapy with cholesterol synthesis enzyme inhibitors or anticipated initiation of such a therapy.
* History of autoimmune disease.
* History of cancer in the last 5 years or wasting disease.
* Intake of prohibited concomitant medication.
* Has known hypersensitivity/allergy to the study drugs.
* Has drug addiction and/or extensive use of alcohol.
* Psychological and/or emotional problems which would render the informed consent invalid or limit the ability of the patient to comply with the study requirements.
* Participation in a clinical investigation within 30 days prior to enrolment in this trial.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2006-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The change from Baseline in Blood pressure (mean reduction in Diastolic Blood Pressure measured at trough). | End of Treatment

SECONDARY OUTCOMES:
The change from Baseline in Adiponectin. | At Final Visit.
The change from Baseline in high sensitivity C-Reactive Protein. | At Final Visit.
The change from Baseline in Fasting Plasma Glucose. | At Final Visit.
The change from Baseline in Fasting Plasma Insulin. | At Final Visit.
The change from Baseline in Insulin Resistance (assessed by Homeostasis Model Assessment Insulin Resistance). | At Final Visit.
The change from Baseline in Lipid Parameters (total cholesterol, low-density lipoprotein cholesterol, high density lipoprotein cholesterol and triglycerides). | At Final Visit.
The change from Baseline in Fibrinogen. | At Final Visit.
The change from Baseline in Prospective Cardiovascular Münster risk score for the assessment of coronary heart disease. | At Final Visit.
The change from Baseline in 24-hour mean blood pressure as assessed by Ambulatory Blood Pressure Measurement. | At Final Visit.
The change from Baseline in Daytime and night-time mean blood pressure Ambulatory Blood Pressure Measurement. | At Final Visit.
The change from Baseline in Systolic Blood Pressure. | End of Treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda Pharma Gmbh, Aachen (Germany)
Locations (24):
- Germany (24):
  - Bad Dürrheim, Baden-Wurttemberg
  - Balingen, Baden-Wurttemberg
  - Deggingen, Baden-Wurttemberg
  - Rottweil, Baden-Wurttemberg
  - Spaichingen, Baden-Wurttemberg
  - Ingolstadt, Bavaria
  - München, Bavaria
  - Passau, Bavaria
  - Schauenburg, Hesse
  - Bocholt, North Rhine-Westphalia
  - Cologne, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Isselburg, North Rhine-Westphalia
  - Roetgen, North Rhine-Westphalia
  - Troisdorf, North Rhine-Westphalia
  - Wesseling, North Rhine-Westphalia
  - Rödersheim-Gronau, Rhineland-Palatinate
  - Dresden, Saxony
  - Freital, Saxony
  - Machem, Saxony
  - Markkleeberg, Saxony
  - Wermsdorf, Saxony
  - Bad Segeberg, Schleswig-Holstein
  - Berlin, State of Berlin